CLINICAL TRIAL: NCT05605678
Title: A Global, Non-interventional Study to Prospectively Evaluate Bleeding Episodes and Treatment Use in Patients with Hemophilia
Brief Title: Hemophilia Non-Interventional Study Prior to SerpinPC Intervention (PRESent-5)
Status: Terminated | Type: Observational
Why Stopped: Study terminated due to business and strategic decision
Sponsor: ApcinteX Ltd (Industry)
Collaborators: Centessa Pharmaceuticals plc (Industry)
Responsible Party: Sponsor
Other Study IDs: AP-0105 (PRESent-5)
Record Dates: First submitted 2022-10-31; First posted 2022-11-04 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Hemophilia a; Hemophilia B
Keywords: Hemophilia; Prospective
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- All Eligible Participants: All Participants diagnosed with severe HemA with or without inhibitors, moderately severe to severe HemB, or HemB with inhibitors will be enrolled and continue to receive their usual hemophilia treatment regimen under SOC therapy. Bleeding episodes and treatment data will be collected during the prospective follow up period in a diary. No intervention will be administered as part of this study.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is a non-interventional study.

SUMMARY:
The primary objective of this study is to obtain prospective baseline documentation of annualized bleeding rates (ABRs) and treatment under standard-of-care (SOC) therapy among participants with hemophilia A or B. Participants in the study may be eligible to enroll in future planned interventional studies to be conducted by Sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Male participants greater than or equal to (>=) 12 and less than or equal to (<=) 65 years of age
2. Who are capable of providing written informed consent (adolescent assent and parental/guardian consent when appropriate) for participation after reading the information and consent form and having the opportunity to discuss the study with the Investigator or their designee
3. With historically documented severe HemA (defined as factor VIII [FVIII] less than (<) 0.01 International Units per milliliter (IU/mL) [<1 percent {%}]), with or without inhibitors, or moderately severe to severe HemB (defined as factor IX [FIX] <=0.02 IU/mL [<=2%]) without inhibitors. Participants must be currently included in a prophylactic treatment program or if undergoing an on-demand treatment regimen must have had >=6 documented acute bleeding episodes (spontaneous or traumatic) that required coagulation factor infusion during the 6 months before enrollment OR: Historically documented HemB (defined as FIX <=0.05 IU/mL [<=5%]) with inhibitors with a historical or ongoing high titer inhibitor [>=5 Bethesda Units/mL] based on medical records or laboratory reports) and an ABR of >=6 in the 6 months before enrollment
4. Who are able to use a diary to document bleeding events and associated treatment

Exclusion Criteria:

1. With known thrombophilia
2. With body weight greater than (>)150 kilogram (kg) or body mass index >40
3. With known current inadequate hematologic function (eg, platelet count <100,000 per microliter [/mcL] and/or hemoglobin level <10 grams per deciliter [g/dL], <100 g/L), hepatic function (that is, total bilirubin >1.5*upper limit of normal [ULN] [excluding Gilbert syndrome], aspartate transferase and/or alanine aminotransferase levels >3*ULN; clinical signs or known laboratory or radiographic evidence consistent with cirrhosis of the liver) or renal function (that is, serum creatinine >2*ULN; based on medical records or available laboratory reports)
4. With previous deep vein thrombosis and pulmonary embolism, myocardial infarction, or stroke
5. With history of intolerance to subcutaneous injections
6. With known current uncontrolled hypertension (systolic blood pressure >160 millimeter of mercury (mm Hg); diastolic blood pressure >100 mm Hg; based on medical records)
7. With active cancer or requires therapy for cancer, except for basal cell carcinoma
8. With concurrent participation in an interventional clinical trial
9. With current or planned use of emicizumab
10. With prior, ongoing, or planned treatment with gene therapy for hemophilia
11. With history of or other evidence of recent alcohol or drug abuse as determined by the Investigator or their designee (in the 12 months before enrollment)
12. With known Human Immunodeficiency Virus (HIV) infection with CD4 count (or T-cell count) of <200 cells/mcL within 24 weeks before enrollment
13. With current or planned treatment with anticoagulant or antiplatelet drugs
14. With any other significant conditions or comorbidities that, in the opinion of the Investigator or their designee, would make the participant unsuitable for enrollment

Ages: 12 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with severe HemA with or without inhibitors, or moderately severe to severe HemB without inhibitors or HemB with inhibitors treated with SOC on-demand or prophylactic hemophilia therapy.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2022-12-09 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2024-11-29 (Actual)

PRIMARY OUTCOMES:
Annualized Bleeding Rate (ABR) for Treated Bleeds and All Bleeds | Minimum 12 weeks
  ABR for treated bleeds and all bleeds at the participant and bleed level (excluding bleeding episodes during surgery and/or procedures).
Average Dose (IU/kg) of Associated Treatment Received for Bleeding Episodes per Hemophilia Product per Time Period and per Bleeding Episode | Minimum 12 weeks

CONTACTS AND LOCATIONS:
Locations (45):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - East Carolina univeristy, Greenville, South Carolina
- Centre of Haematology named after prof. R. O. Yeolian, Yerevan, Yerevan, Armenia
- Royal Prince Alfred Hospital, Camperdown, Camperdown, Australia
- Brazil (2):
  - Fundacao de Desenvolvimento da Unicamp FUNCAMP, Campina, São Paulo
  - HEMOES - Centro de Hemoterapia e Hematologia do ES, Vitória, Vitória
- Canada (3):
  - Hamilton Health Sciences Corporation, Hamilton, Hamilton
  - Hamilton Health Sciences Corporation, Hamilton, Ontario
  - Unity Health Toronto, Toronto, Toronto
- Ain Shams University, Cairo, Cairo Governorate, Egypt
- France (4):
  - Hopital Necker - Enfants Malades, Paris, Paris
  - Hospices Civils de Lyon (HCL) - Hopital Femme-Mere-Enfant (HFME), Lyon, Rhone
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - CHU Hotel Dieu, Nantes
- Germany (3):
  - University Hospital Frankfurt, Frankfurt am Main, Hesse
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden, Saxony
  - Klinik fur Angiologie Hamostaseologie Haus 12 A Gerinnungssprechstunde, Berlin, State of Berlin
- India (3):
  - St. Johns Medical College, Bangalore, Bangalore
  - K J Somaiya Super Speciality Hospital & Research Centre, Mumbai, Mumbai
  - Christian Medical College & Hospital, Ludhiana, Punjab
- Italy (2):
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan, Milano
  - Azienda Ospedaliero-Universitaria Careggi, Florence
- Poland (2):
  - Korczowski Bartosz, Gabinet Lekarski, Rzeszów, Podkarpackie Voivodeship
  - Kl Hemat Now Krwi i Trans USK, Wroclaw, Wrocław
- South Africa (2):
  - King Edward VIII Hospital, Durban, Durban
  - Phoenix Pharma (Pty) Ltd, Port Elizabeth, Eastern Cape
- Spain (4):
  - Hospital Regional Universitario de Malaga Hospital Carlos Haya - Hospital Materno-Infantil, Málaga, Malaga
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia, Murcia
  - Hospital Universitario Miguel Servet, Zaragoza, Zaragoza
  - Hospital Universitari Vall d'Hebron, Barcelona
- Taiwan (4):
  - China Medical University Hospital, Taichung, Taichung
  - Chung Shan Medical University, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
- Turkey (Türkiye) (2):
  - Ege University Hospital, Izmir, İzmir
  - Ege University Medical Faculty Pediatric Hospital, Izmir
- United Kingdom (9):
  - University Hospital of Wales, Cardiff, Cardiff
  - Glasgow Royal Infirmary, Glasgow, Glasgow
  - Barts and London School of Medicine and Dentistry, London, London
  - Royal Free London NHS Foundation Trust, London, London
  - Imperial College Healthcare NHS Trust, London, London
  - Southampton General Hospital, Southampton, Southampton
  - Royal Victoria Infirmary, Newcastle upon Tyne, Tyne and Wear
  - Kent Canterbury Hospital, Canterbury
  - Central Manchester University Hospitals NHS Foundation Trust - Manchester Royal Infirmary, Manchester

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD due to the Sponsor's strategic and data-driven decision to discontinue the global clinical development of SerpinPC.